CLINICAL TRIAL: NCT03459989
Title: Accuracy of Two Dimensions Ultrasonography of Fetal Thigh Soft Tissue Versus Hadlock's Formula in Estimation of Fetal Weight
Brief Title: Comparison Between Fetal Thigh Soft Tissue Versus Hadlock's Formula in Estimation of Fetal Weight by Ultrasound
Acronym: STT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed abd elfatah elsenity, Lecturer, Ain Shams University
Other Study IDs: 9071729
Record Dates: First submitted 2018-03-04; First posted 2018-03-09 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Estimation of Fetal Weight
Keywords: hadlock; thigh soft tissue
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- pregnant women: we will measure expected fetal weight by ultrasound by hadlock's formula and thigh soft tissue for each pregnant woman
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Samsung H60 Ultrasound

SUMMARY:
We are going to do 2d ultrasound to compare between hadlock's formula and thigh soft tissue formula in expecting the after birth fetal weight and to find which of these formulas to be more accurate

DETAILED DESCRIPTION:
We are going to do 2d ultrasound to 200 pregnant women between 38 weeks to 40 weeks singleton pregnancy in Ain Shams University Maternity Hospital to measure the expected fetal weight by hadlock's formula and thigh soft tissue formula and then we are going to measure the actual fetal weight after birth of these 200 fetuses and to find out which formula to be more accurate in estimation of fetal weight

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age 38 - 40 wks
2. Singleton uncomplicated pregnancies
3. Normal amniotic fluid volume

Exclusion Criteria:

Women with one of the following conditions:

1. Fetuses with congenital anomalies,
2. The biometric measurements of those, which were unable to ascertain due to reasons like deeply engaged head, very thick abdominal wall etc.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women between 38 weeks and 40 weeks
Study Population: The study population comprises 200 pregnant women at 38 to 40 week of gestation attending outpatient clinic and emergency Ain Shams University Maternity Hospital, Obstetrics and Gynaecology Department, Faculty of medicine.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-10-30 (Estimated)

PRIMARY OUTCOMES:
Fetal weight | 38 weeks to 40 weeks of gestation
  hadlock's 4th formula and thigh soft tissue formula

CONTACTS AND LOCATIONS:
Overall Officials: Adel SH Salah El-Din, Professor, Study Chair — Ain Shams University
Locations (1):
- Ain Shams Universitiy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided